CLINICAL TRIAL: NCT05779267
Title: NRX-101 for Treatment-Resistant Bipolar Depression in Patients At Risk for Self-Harm
Brief Title: NRX-101 Expanded Access
Acronym: NRX-101EAP
Status: Available | Type: Expanded Access
Sponsor: NeuroRx, Inc. (Industry)
Collaborators: Prevail Infoworks (Industry)
Responsible Party: Sponsor
Other Study IDs: NRX-101_006 EAP
Record Dates: First submitted 2023-03-08; First posted 2023-03-22 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Bipolar Depression; Bipolar Affective Disorder
Keywords: bipolar depression; suicidal ideation; cycloserine; NMDA antagonist; NRX-101
MeSH Terms: conditions — Bipolar Disorder; Suicidal Ideation

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: NRX-101 — D-cycloserine/lurasidone fixed dose combination

SUMMARY:
There is no currently-approved pharmacotherapy for patients with Treatment-Resistant Bipolar Depression and Suicidal Ideation or behavior. The purpose of this Expanded Access Treatment Protocol is to make NRX-101 available to patients who have depression and suicidal ideation despite treatment with currently approved medication and to gather information on safety and efficacy in a real-world data environment. Participants will be treated by their own practicing psychiatrist and will agree to periodic psychometric evaluations to assess depression, suicidal ideation, and side effects.

DETAILED DESCRIPTION:
INTRODUCTION

1 Suicidal Ideation and Behavior in Bipolar Disorder

Bipolar Disorder (formerly known as manic depressive disorder) is a well-established psychiatric diagnosis, with a prevalence of about 2.6% in the United States (approximately 8.5 million people) (Kessler et al., 2005). The risk of subacute suicidal ideation or behavior (SSIB) is uniquely high in patients during bipolar depressive episodes, compared to those with major depressive disorder (MDD), thought disorders, and personality disorders. Lifetime suicide behavior occurs in 25% to 56% of people with bipolar disorder (Nierenberg et al., 2001). About 40% of the nearly 50,000 annual deaths from suicide in the United States are associated with bipolar disorder (Mahli et al., 2015). The overall rate of death by suicide among patients with bipolar disorder is 164 per 100,000 person-years, compared to about 14 per 100,000 person-years for the general population. Those who have attempted suicide are 2.3 times more likely to die by suicide compared to those without a suicide attempt (Coryell et al., 2016). Thus, bipolar depression with suicidal ideation has uniquely lethal clinical characteristics (Pompili, et al., 2013).

6.2 Current Treatment Options

Despite its lethal characteristics, there is no approved pharmacologic treatment for patients with bipolar depression and suicidal ideation. Electroconvulsive therapy (ECT), often combined with inpatient psychiatric care, remains the only Food and Drug Administration (FDA)-approved treatment for patients with acute suicidal ideation in bipolar depression, despite ECT's well-documented side effects that include memory loss and confusion, along with its high cost. However, the toxicity of ECT is such that it is less likely to be used in patients with subacute levels of suicidal ideation and no oral medication has been shown to reduce suicidal ideation in patients with depression in general or bipolar depression in specific. Physicians are increasingly cautious about the use of selective serotonin release inhibitors (SSRIs), particularly in patients with suicidal ideation because of evidence that SSRIs and other antidepressants may actually increase the risk of suicidal ideation, particularly in younger patients (Stone et al., 2009). This evidence has resulted in an FDA warning on the label of current antidepressants. Moreover, it seems clear that antidepressants do not decrease SSIB in proportion to their mitigating effect on symptoms of depression.

In recent years, several combined D2/5-HT2A antagonists have shown efficacy in treating bipolar depression (olanzapine/fluoxetine combination, quetiapine, and lurasidone) with treatment guidelines endorsing common use as first-line standard of care treatment in acute bipolar depression. While these medications are effective at reducing overall symptoms of depression, they do not specifically reduce suicidal ideation, as shown in recent clinical trials of lurasidone (Loebel et al., 2014a; Loebel et al., 2014b). Moreover, in these two studies, individuals with active suicidal ideation (Montgomery Asberg Depression Rating Scale [MADRS] item 10 ≥ 4) were specifically excluded because of concerns regarding the possibility of exacerbating suicidality with these medications. Similarly, acutely suicidal patients are routinely excluded from clinical trials of other experimental anti-depressive agents. Thus, bipolar depression with suicidal ideation represents a major unmet medical need that must frequently be treated with voluntary or involuntary hospitalization under highly supervised conditions and ECT.

6.3 Preclinical Models of Anxiety and Akathisia

Although the mechanisms mediating antidepressant-related increases in suicide remain unclear, leading theories suggest that increases in anxiety/akathisia may play a critical role (Harada et al., 2014; Popovic et al., 2015). Serotonin-related anxiety/akathisia may be modeled in rodents using several well-established assay systems, such as the elevated plus maze, and are known to be sensitive to serotonergic agents (Sachdev and Brune, 2000). In this assay, reduced percent time spent in the open arms of the maze is believed to be associated with increased akathisia and anxiety. In contrast, increased total distance traveled in the maze is thought to be a signal related to psychosis. As shown by Javitt (2014), D-cycloserine (DCS) significantly reduces the anxiogenic effects of lurasidone and quetiapine, as measured by time spent in open arms, suggesting that this treatment might reduce medication-induced suicidality, as well as suicidality associated with bipolar depression itself.

Preclinical data, using the Rodent Akathisia model, suggests a potential synergistic interaction between DCS and lurasidone. On one hand, as described above, DCS appears to block the anxiogenic effects of lurasidone. On the other hand, lurasidone may reverse the low-level psychotomimetic effects of DCS. Lurasidone mediates its antipsychotic effects at both D2 and 5-HT2A receptors. As opposed to pure serotonergic agents used in the treatment of major depressive disorders (e.g., SSRIs), the additional D2 blockade of lurasidone makes it a clinically effective antipsychotic; thus, it could also be effective in treating the psychotic symptoms that may be induced by an N-methyl-D-aspartate receptor (NMDAR) antagonist.

Clearly, the phenomena observed in rodents should not be viewed as isomorphic with drug-induced akathisia and/or restlessness/anxiety syndrome in humans. However, these findings provide a rationale for combining glycine site-binding NMDAR antagonists with 5-HT2A antagonists in phase 2 and 3 studies of otherwise-safe drugs for the treatment of bipolar depression. This is particularly true in situations where akathisia is believed to predispose vulnerable patients to suicide.

6.4 Clinical Experience with DCS

Antidepressant effects of high-dose DCS were first noted in the late 1950s when it was introduced as a treatment for tuberculosis (TB). Several clinicians noted a dramatic improvement in patients' depressive symptoms, leading to suggestions of DCS' potential psychotropic effects. These effects were subsequently confirmed in small-scale clinical studies (Crane, 1959 and 1961). The mechanism of action was unknown at the time, and the finding was not pursued. The interaction of DCS with the NMDAR was first demonstrated in 1989 (Hood et al., 1989), leading to some interest in NMDAR blockers as potential antidepressant treatments (Trullas and Skolnick, 1990; Skolnick et al., 1996). For example, both DCS and the related compound aminocyclopropanecarboxylic acid (ACPC) were shown to be active in mice, using the forced swim test for depression (Lopes et al., 1997). To the best of our knowledge, no clinical antidepressant research programs targeting the NMDA receptor were initiated at that time.

Interest in the potential clinical use of DCS as an antidepressant agent was renewed following Berman's fortuitous observation of ketamine's rapid antidepressant effect (Berman et al., 2000). An initial study performed with DCS at a dose of 250 mg/day did not show therapeutic effects, but it did demonstrate a relative lack of psychotomimetic side effect when DCS was combined with concurrent antidepressant treatment (Heresco-Levy et al., 2006). Based upon these safety data, a study using a higher dose of 1000 mg/day was initiated, with results reported in 2013 (Heresco-Levy et al., 2013). At the higher dose of 1000 mg/day, significant beneficial effects were observed in 13 subjects vs. placebo control with SSRI-nonresponsive depressive symptoms. The improvements were manifested within 2 weeks and persisted throughout the 6-week treatment period. These data suggest a >0.9 effect size. In that study, a slow DCS titration was used, with 250 mg/day for 3 days, followed by 500 mg/day for 18 days (i.e., until the end of week 3); followed by 750 mg/day for 1 week (i.e., until the end of week 4), followed by 1000 mg/day (i.e., until the end of study). A statistically significant improvement was observed in the DCS group compared to placebo by the end of week 4, i.e., within 1 week of initiation of a DCS dose >500 mg/day

The phase 2 STABIL-B trial provides evidence of efficacy from a study of NRX-101 versus Lurasidone in patients with severe bipolar depression (MADRS ≥ 30) and Acute Suicidal Ideation or behavior (C-SSRS 4, or 5), after initial stabilization with a single infusion of ketamine.

6.5 Investigational Therapy Following screening and informed consent, participants will be treated with NRX-101 twice daily by mouth. It is anticipated that participants will also be receiving concurrent bipolar disorder-directed treatment with various predefined combinations of medications. This treatment regimen will be maintained upon entry into the study. However, any use of lurasidone, quetiapine, aripiprazole, risperidone, brexpiprazole, olanzapine, cariprazine, or lumateperone, will be discontinued at study entry because NRX-101 contains a therapeutic dose of lurasidone. The treating psychiatrist should ensure that any medications to be discontinued can be done so safely. At entry, at the discretion of the investigators or the delegated treating physician subjects may continue their mood stabilizers which should not change over the course of the trial. In addition, participants receiving the olanzapine/fluoxetine combination will continue to receive the fluoxetine component.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years of age, inclusive, at Screening
2. Able to understand and provide written and dated informed consent prior to screening
3. Deemed likely to comply with the study protocol, including communication of adverse events (AEs) and other clinically important information, including adherence to the text messaging component of the trial.
4. Will follow medical directions for psychiatric care, as appropriate, per the standard of care.
5. Resides in a stable living situation. A stable living situation will be defined as a minimum of 3 months at the same address with a reasonable expectation that the situation will continue such that the patient's ability to participate in the study will not be affected. Please note that housing in a shelter of any kind will not be deemed stable housing.
6. Must have been under the care of a licensed qualified psychiatric prescriber for a minimum of 6 months prior to screening and be able and willing to provide documentation of treatment history and current and past psychiatric medication.
7. Has an identified reliable informant/care partner, that is willing to provide information and/or supportive care as necessary.
8. Diagnosed with bipolar disorder (BD) I or II according to the criteria defined in the DSM-5. The diagnosis of BD will be made by a psychiatrist or other qualified licensed psychiatric provider able to render a diagnosis and be supported by the MINI 7.0.2.
9. Confirmed active suicidal ideation (without the intention to act) as evidenced by an answer of 'Yes' on item 3 and/or 4 and not requiring hospitalization at Screening and an answer of 'No' on item 5 of the C-SSRS within 4-weeks of Screening
10. A total score greater than or equal to 20 on the 10 items of the MADRS
11. No co-morbidities, as ascertained by medical history clinical laboratory evaluations, and electrocardiogram (ECG) which might interfere with compliance or the ability to assess efficacy or safety.
12. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following criteria, and agrees to continue use of the same method of birth control for the duration of study participation:

    1. Non-childbearing potential: physiologically incapable of becoming pregnant (i.e. permanently sterilized [status post-hysterectomy, bilateral tubal ligation] or post-menopausal with last menses at least one year prior to screening); or
    2. Childbearing potential, and meets the following criteria:

    i. Use of any form of hormonal birth control for at least 2 months prior to Screening, on hormone replacement therapy that started prior to 12 months of amenorrhea, using an intrauterine device (IUD) for at least 1 month prior to Screening, in a monogamous relationship with a partner who has had a vasectomy, or sexually abstinent.

    ii. Negative urine pregnancy test at Screening, confirmed by a second negative urinary pregnancy test at Day 1, prior to receiving any study treatment
13. Body mass index (BMI) between 18-40 kg/m2.
14. If receiving concurrent psychotherapy, the type and frequency of the therapy (e.g., weekly or monthly) has been stable for at least 3 months prior to Screening and is expected to remain stable for the duration of study participation
15. Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, benzodiazepines, maximum 2mg/daily, or trazodone) will be allowed if the therapy has been stable for at least 4-weeks prior to screening and if it is expected to remain stable during the course of the patient's participation in the study. Participants can also continue treatment with benzodiazepines maximum dose 2mg/daily used for anxiety if therapy has been stable relative to dose and schedule for at least 4-weeks prior to screening and if it is expected to remain stable during the course of the patient's participation in the study. If receiving concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, benzodiazepines, or trazodone), the therapy has been stable for at least 4 weeks prior to Screening and is expected to remain stable for the duration of study participation.
16. If receiving benzodiazepines for anxiety, the dose and frequency have been stable for at least 4 weeks prior to Screening and is expected to remain stable for the duration of study participation
17. If women are receiving hormone replacement therapy or estrogen replacement, the therapy has been stable for at least 3 months prior to Screening and is expected to remain stable for the duration of study participation

Exclusion Criteria:

* 1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.

  2. Female who is pregnant or breastfeeding. 3. Female with a positive pregnancy test at Screening or prior to randomization.

  4. Current DSM-5 diagnosis of moderate or severe substance use or abuse disorder or a diagnosis of dependence (except marijuana or tobacco use disorder only) within the 12 months prior to Screening. (Note: Substance abuse cannot be the precipitant for study entry.) 5. A lifetime history of
  1. phencyclidine (PCP)/ketamine drug abuse, or
  2. failed use of ketamine for depression or suicidality. 6. History of schizophrenia or schizoaffective disorder, or any history of psychotic symptoms when not in an acute bipolar mood episode.

     7. History of anorexia nervosa, bulimia nervosa, eating disorder not otherwise specified (NOS), or other specified feeding and eating disorders (OSFED) within 5 years of Screening.

     8. Has dementia, delirium, amnestic, or any other cognitive disorder. 9. Current major psychiatric disorder, diagnosed at Screening with the MINI 7.0.2 which is the primary focus of treatment, with bipolar disorder as the secondary focus of treatment, within the past 6 months.

     10. Estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73 m2 using the Cockcroft-Gault formula 11. A clinically significant abnormality on the Screening physical examination that may affect safety or study participation, or that may confound interpretation of study results according to the study clinician.

     12. Current episode of:

  a. Myocardial infarction within 1 year of Screening. b. Diagnosis of angina pectoris. c. Prolonged QTc interval, as measured by Fridericia's correction formula (QTcF) ≥450 msec at Screening for males or ≥ 470 msec for females on 2 of 3 measurements at least 15 minutes apart prior to randomization on Day 1.

  13. Diagnosis of chronic lung disease, excluding asthma. 14. Lifetime history of any of the following: surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's Disease, Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention that, according to the clinician, is deemed associated with significant injury to, or malfunction of, the CNS.

  15. History of significant head trauma within the past two years. 16. Diabetes mellitus fulfilling any of the following criteria:
  1. Unstable diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >8.0 % at Screening.
  2. Admitted to the hospital for treatment of diabetes mellitus or diabetes mellitus-related illness in the past 12 weeks.
  3. Not under physician care for diabetes mellitus.
  4. Not on the same dose of oral hypoglycemic drug(s) and/or diet for the 4 weeks prior to Screening.
  5. Not on the same dose of oral thiazolidinediones (glitazones) for the 8 weeks prior to Screening.

     17. Any current or past history of any physical condition which, in the opinion of the investigator, may put the patient at risk or interfere with study results interpretation.

     18. Diagnosis of HIV/AIDS 19. Diagnosis of Hepatitis C 20. On exclusionary concomitant psychotropic and non-psychotropic medications (see Appendix 1).

     21. Prescribed more than one agent in each of the following categories at randomization:

  <!-- -->

  1. Approved SSRIs
  2. Approved serotonin and norepinephrine reuptake inhibitors (SNRIs)
  3. Approved tetracyclic antidepressants (TeCAs)
  4. Approved Mood stabilizers (e.g. lithium, valproic acid, and lamotrigine) Note: Any/all 5hT2A medications will be discontinued at study entry. Participants currently on Lurasidone will be randomized to either standard of care or NRXx-101 at the indicated starting dose 22. Currently prescribed oxcarbazepine or carbamazepine 23. Exclusionary laboratory values or any other clinically significant abnormal laboratory result (as determined by the investigator and Medical Monitor) at Screening.

     24. Known allergies to lurasidone or Latuda®, cycloserine or Seromycin®, or the following excipients: mannitol, croscarmellose sodium, magnesium stearate, silicon dioxide, and/or hydroxypropylmethylcellulose (HPMC).

     25. Participation in any clinical trial with an investigational drug or device within the past month or planned concurrent study participation.

     26. Study site personnel and/or persons employed by NRx Pharma, Inc., the Contract Research Organization (CRO), the investigator, or study site (i.e., permanent, temporary contract worker, or designee responsible for the conduct of the study), or an immediate family member (i.e., spouse, parent, child, or sibling [biological or legally adopted]) of such persons.

     27. Positive urine toxicity screening for use of any cocaine, opiates and non-prescribed amphetamine and non-prescribed barbiturates (Note: Cannabinoids or Marijuana use is not exclusionary unless it meets the DSM-5 criteria for abuse disorder or dependence) 28. Signs and symptoms of active or residual COVID-19, or unresolved symptoms of COVID-19 that impact health, e.g. requirements for oxygen supplementation, etc. Discharge from an inpatient hospitalization for more than 48 hours for COVID-19 within the past 28 days.

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Javitt, MD, MPH, Principal Investigator — NRx Pharmaceuticals; Martin Brecher, MD, Study Director — NRx Pharmaceuticals

REFERENCES:
- See also: NRX-101 (D-cycloserine plus lurasidone) vs. lurasidone for the maintenance of initial stabilization after ketamine in patients with severe bipolar depression with acute suicidal ideation and behavior: A randomized prospective phase 2 trial — https://www.medrxiv.org/content/10.1101/2022.08.11.22278658v1.full